CLINICAL TRIAL: NCT03172533
Title: Prospective, Randomized, Double-blind, Placebo-controlled Clinical Trial on the Effects of an Estrogen-progestin Combination as add-on to Inpatient Psychotherapy in Adult Female Patients Suffering From Anorexia Nervosa
Brief Title: Estrogen Replacement in Anorexia Nervosa
Acronym: HOSAN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties in recruitment
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UKER-AN-HS-01
Record Dates: First submitted 2017-05-22; First posted 2017-06-01 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa; estrogen; psychotherapy; cortisol; appetite regulation; neurocognitive performance; eating disorder; sexual hormone
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders | interventions — Ethinyl Estradiol; dienogest

STUDY DESIGN:
Intervention Model Description: randomized, placebo-controlled Phase IIa clinical trial in patients with anorexia nervosa
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- verum group (Active Comparator): approved oral contraceptive: ethinyl estradiol 0.03mg and dienogest 2mg (combination drug) daily intake over 10 weeks
  Interventions: Drug: ethinyl estradiol 0.03mg and dienogest 2 mg (combination)
- placebo group (Placebo Comparator): placebo
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: ethinyl estradiol 0.03mg and dienogest 2 mg (combination) — approved oral contraceptive (Germany): Maxim
  Arms: verum group
Drug: Placebo oral capsule — placebo
  Arms: placebo group

SUMMARY:
The present study is a placebo-controlled randomised study on the effects of estrogen replacement upon AN-associated psychopathology, several neurocognitive domains and appetite-regulating circuits in female patients with AN.

The investigators aim at assessing peripheral concentrations of neuroendocrinological components of the Hypothalamus-Pituitary-Gonadal (HPG) and Hypothalamus-Pituitary-Adrenal (HPA) axis, as well as appetite-regulating hormones in AN and to examine associations with AN-associated psychopathology and neurocognitive performances before (baseline), during and after inpatient psychotherapy of female patients receiving concomitant treatment with estrogens (vs. placebo).

DETAILED DESCRIPTION:
While there is broad knowledge on the disruption of appetite regulation, neurocognitive deficits in AN patients, the impact of cortisol on neurocognitive performances in patients with AN and the effects of estrogen on neurocognitive features in healthy subjects, up to now, no study has implemented estrogen replacement in AN patients, in order to examine ist effects upon AN-associated psychopathology, neurocognition and peptides regulating appetite. Thus, this is the first study of its kind.

Primary target: Assessment of the impact of sexual hormone replacement using an estrogen-progestin-combination as add-on to psychotherapy upon neurocognitive performance in patients suffering from anorexia nervosa by means of a neuropsychological test battery consisting of a test of verbal intelligence, the Trail making test A and B, a Go/No-go paradigm and the Wisconsin Card Sorting Test.

Secondary targets:

* Examination of safety and tolerability of sexual hormone replacement using an estrogen-progestin-combination in patients with anorexia nervosa.
* Assessment of the impact of the sexual hormone replacement upon psychopathology in patients with anorexia nervosa by means of the Eating Disorder Examination Questionnaire (EDE-Q) and the Eating Disorder Inventory-2 (EDI-2).
* Assessment of the impact of substitution upon anxiety (STAI)
* Assessment of the impact on cortisol levels
* Assessment of the impact on appetite-regulating plasma peptides
* Assessment of the impact on the prescription of antidepressants

ELIGIBILITY:
Inclusion Criteria:

* anorexia nervosa according to the Diagnostic and Statistical Manual of Mental Disorders (DSM V) or subsyndromal anorexia nervosa (lack of a diagnostic symptom according to DSM V)
* BMI ≥ 13 kg/m2 and ≤ 18.5 kg/m2
* able to provide written informed consent

Exclusion Criteria:

* a known hypersensitivity to the active compound or to other components of the study drug
* one or more contraindications for the use of hormonal contraception: Smoking over 20 cigarettes/day; Acute venous thromboembolic disease or increased risk; Known hereditary or acquired predisposition for venous thrombosis, e.g. activated protein C (APC)-resistance (including factor V Leiden Mutation), antithrombin III deficiency, protein C deficiency, protein S deficiency; Risk for arterial thromboembolism (diabetes mellitus with vascular sequelae, severe hypertonus, severe dyslipoproteinemia); Known hereditary or acquired predisposition for arterial thrombosis, e.g. hyperhomocysteinemia and anti-phospholipid antibodies (anticardiolipin antibodies, Lupus anticoagulants); Cerebrovascular disease (past cerebral infarction or prodromal states such as transitory ischemia attacks); Past migraine with focal neurological symptoms; Liver disease or pancreatitis; Dubin-Johnson syndrome and Rotor syndrome; Known porphyria; Known or suspected sexual hormone sensitive tumors; Unresolved vaginal bleeding
* a present severe depressive episode (major depression) according to the DSM V
* past or present alcohol or drug abuse
* severe psychiatric disorders (axis I) according to the DSM V (such as bipolar affective disorder or schizophrenia) in addition to anorexia nervosa
* suicidality
* known diabetes mellitus
* severe somatic comorbidity or organ dysfunction that is not compatible with intake of the study drug
* use of hormonal depot compounds (injectable drugs, implants), or hormonal intrauterine pessaries during the last four weeks before the screening visit (V1)
* pregnancy
* breastfeeding during the last 6 months before V1

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Changes in neurocognitive performance | 10 weeks of hormonal substitution with an estrogen-progestin-combination
  Performance based on a neurocognitive test battery

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse Events (AE) (safety/tolerability) | 10 weeks of hormonal substitution with an estrogen-progestin-combination
  Number of adverse events (including AE, AR, severe AE, SAR and SUSAR)
Changes in psychopathology (EDE-Q) | 10 weeks of hormonal substitution with an estrogen-progestin-combination
  Changes in sum scores in the EDE-Q
Changes in psychopathology (EDI-2) | 10 weeks of hormonal substitution with an estrogen-progestin-combination
  Changes in sum scores in the EDI-2
Changes in psychopathology (STAI) | 10 weeks of hormonal substitution with an estrogen-progestin-combination
  Changes in sum scores in the STAI
Changes in psychopathology (Patient Health Questionnaire-9, PHQ-9) | 10 weeks of hormonal substitution with an estrogen-progestin-combination
  Changes in sum scores in the PHQ-9
Changes in psychopathology (Eating Disorder Quality of Life, EDQoL) | 10 weeks of hormonal substitution with an estrogen-progestin-combination
  Changes in sum scores in the EDQoL
Neuroendocrinological changes (cortisol) | 10 weeks of hormonal substitution with an estrogen-progestin-combination
  Changes in plasma cortisol levels during a dexamethasone suppression test
Neuroendocrinological changes (glucose) | 10 weeks of hormonal substitution with an estrogen-progestin-combination
  Changes in plasma concentrations of glucose
Neuroendocrinological changes (insulin) | 10 weeks of hormonal substitution with an estrogen-progestin-combination
  Changes in plasma concentrations of insulin
Neuroendocrinological changes (ghrelin) | 10 weeks of hormonal substitution with an estrogen-progestin-combination
  Changes in plasma concentrations of the appetite-regulating peptide ghrelin
Neuroendocrinological changes (leptin) | 10 weeks of hormonal substitution with an estrogen-progestin-combination
  Changes in plasma concentrations of the appetite-regulating peptide leptin
Changes in antidepressant medication | 10 weeks of hormonal substitution with an estrogen-progestin-combination
  Changes in antidepressants´ use

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychosomatic Medicine and Psychotherapy, University Hospital Erlangen, Erlangen, Bavaria, Germany

REFERENCES:
- [Derived] Paslakis G, Maas S, Gebhardt B, Mayr A, Rauh M, Erim Y. Prospective, randomized, double-blind, placebo-controlled phase IIa clinical trial on the effects of an estrogen-progestin combination as add-on to inpatient psychotherapy in adult female patients suffering from anorexia nervosa. BMC Psychiatry. 2018 Apr 10;18(1):93. doi: 10.1186/s12888-018-1683-1. PMID 29631553